CLINICAL TRIAL: NCT05766306
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Study Investigating the Efficacy of a Probiotic Blend on Stress in Adolescents With Moderate Perceived Stress
Brief Title: The Efficacy of a Probiotic Blend on Stress in Moderately Stressed Teens
Acronym: TEEN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lallemand Health Solutions (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: L-024
Record Dates: First submitted 2023-02-09; First posted 2023-03-13 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2023-08

CONDITIONS: Stress
Keywords: probiotics; probiotic; stress; adolescents; teenagers; teens

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double-blinded.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Participants will be randomized to receive the probiotic blend for 56 days.
  Interventions: Dietary Supplement: Probiotic Blend
- Placebo (Placebo Comparator): Participants will be randomized to receive the placebo for 56 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic Blend — Participants will be taking 1 sachet a day, 3 billion CFU.
  Arms: Probiotic
Dietary Supplement: Placebo — Participants will be taking 1 sachet a day.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to test to efficacy of a probiotic blend on stress in adolescents with moderate perceived stress. It is hypothesized that those taking the probiotic blend will have decreased levels of stress compared to those receiving the placebo.

DETAILED DESCRIPTION:
Participants in this randomized, double-blind, placebo-controlled, parallel study will be adolescents with moderate perceived stress. Participants will be enrolled in this study for 63 days, with a 56-day intervention period and a 7 day follow-up period. There will be a total of 5 visits: 4 in-person and 1 follow-up phone call.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 13 and 17 years, inclusive
2. Individuals of child-bearing potential must have a negative screening urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:

   * Abstinence or agrees to use contraception if planning to become sexually active
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner at least 6 months prior to screening
3. Enrolled in and currently attending school at baseline and for the duration of the study period
4. Individuals with moderate stress as determined by a score of 14-26 on the PSS
5. Does not have an anxiety disorder as determined by QI assessment of the YAM-5
6. Can fluently read and speak English
7. Willing to discontinue consumption of probiotic supplements, probiotic fortified products (e.g., fortified yogurt) and fiber supplements (e.g., Metamucil, Benefiber) for the corresponding washout period indicated in Section 7.3.2 and throughout the study
8. Willingness to maintain current lifestyle habits as much as possible throughout the study including diet, exercise, sleep, and non-pharmacological therapies (e.g., meditation, yoga, breathing exercises)
9. Willingness and ability to complete questionnaires, records and diaries associated with the study and to complete all clinic visits
10. Willingness to provide biological samples (saliva, urine, stool) three times during the study
11. The child and the child's parent(s) or legal guardian(s) to provide voluntary, written, informed assent and consent, respectively, for their child to participate in the study
12. Healthy as determined by medical history as assessed by Q

Exclusion Criteria:

1. Individuals who are pregnant, breast feeding, or planning to become pregnant during the study
2. Allergy, sensitivity, or intolerance to the investigational product or placebo ingredients
3. Previous diagnosis or treatment of a mental health disorder or neurodevelopmental disorder, including anxiety disorders (e.g., generalized anxiety disorder, post-traumatic stress disorder, obsessive compulsive disorder, seasonal affective disorder), mood disorders (e.g., major depressive disorder, bipolar disorder) or attention deficit/hyperactivity disorder within the last two years as assessed by the QI
4. Current diagnosis of a sleep disorder (e.g., obstructive sleep apnea, sleep terrors, parasomnia, restless leg syndrome), or a disorder which requires medication that may affect sleep as assessed by the QI
5. Previous diagnosis of neurological diseases (e.g., epilepsy, muscular dystrophy, cerebral palsy) assessed by the QI
6. Currently suffering from periodontitis as assessed by the QI
7. Travelled across 1 or more time zones in the last 3 weeks prior to baseline and/or is anticipating more travel during the study period
8. Current or history of any significant diseases of the gastrointestinal tract (e.g., Crohn's disease, ulcerative colitis, peptic ulcer disease) as assessed by the QI
9. Individuals with an autoimmune disease or are immune compromised
10. Use of medical cannabinoid products as assessed by the QI
11. Use of cannabinoid, tobacco or nicotine-containing products, or alcohol consumption
12. Alcohol or drug abuse within the last 12 months
13. Regular consumption of over-the-counter medications, supplements (e.g., melatonin), foods or drinks that may affect stress or sleep. The participant may be eligible after a washout period prior to their baseline visit and if they agree to discontinue use of the product throughout the study.
14. Current use of prescribed medications that may affect stress, sleep and/or mood
15. Current use of antibiotics. The participant may be eligible after a 30-day washout period prior to their baseline visit
16. Participation in other clinical research studies 30 days prior to baseline, as assessed by the QI
17. Individuals who are cognitively impaired and/or unable to give informed consent
18. Any other condition or lifestyle factor, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
Change in stress at day 56 from baseline | 56 days
  The difference in change from baseline in stress at Day 56 between Probiotic and Placebo measured by the Perceived Stress Scale (PSS).
  The PSS is a validated and commonly used tool to measure perceived stress. Responses are rated by participants on a 5-point Likert scale. The PSS-10 has been reported to be superior to other versions of the scale and will be used in this study. The total score of PSS-10 ranges between 0-40. Scores between 0-13 are considered low stress, 14-26 are considered moderate stress, and 27-40 are considered high stress.

SECONDARY OUTCOMES:
Change in stress at day 28 from baseline | 28 days
  The difference in change from baseline in stress at Day 28 between Probiotic and Placebo measured by the Perceived Stress Scale (PSS) The PSS is a validated and commonly used tool to measure perceived stress. Responses are rated by participants on a 5-point Likert scale. The PSS-10 has been reported to be superior to other versions of the scale and will be used in this study. The total score of PSS-10 ranges between 0-40. Scores between 0-13 are considered low stress, 14-26 are considered moderate stress, and 27-40 are considered high stress.
Change in sleep quality from baseline | 56 days
  The difference in change from baseline at Days 28 and 56 between Probiotic and Placebo in sleep quality as assessed by the Adolescent Sleep-Wake Scale (ASWS).
  The ASWS is a 28-item scale developed to assess self-reported sleep quality in individuals 12-18 years old. The scale is comprised of five behavioral dimensions including going to bed (5 questions), falling asleep (6 questions), maintaining sleep (6 questions), reinitiating sleep (6 questions), and returning to wakefulness (5 questions). Respondents are instructed to provide responses based on the past month on a six-point Likert scale ranging from always (score=1) to never (score=6). Higher scores representing better sleep quality.
Change in daytime sleepiness from baseline | 56 days
  The difference in change from baseline at Day 28 and 56 between Probiotic and Placebo in daytime sleepiness as assessed by the Cleveland Adolescent Sleepiness Questionnaire (CASQ) The CASQ is a tool developed to assess daytime sleepiness among adolescents aged 11-17 years old. The questionnaire is a self-reported tool comprised of 16 questions with responses ranging from "Never (0 times per month)" to "Almost every day (5 or more times per week)" and respondents are instructed to indicate their response that best represents how often it applies to them . Higher scores represent greater sleepiness.
Change in sleep-related hormones from baseline | 56 days
  The difference in change from baseline at Days 28 and 56 between Probiotic and Placebo in sleep-related hormones as assessed by morning salivary cortisol, and nighttime salivary melatonin
Change in stress-related hormones from baseline | 56 days
  The difference in change from baseline at Days 28 and 56 between Probiotic and Placebo in stress-related hormone as assessed by urinary free cortisol
Change in mood from baseline | 56 days
  The difference in change from baseline at Days 28 and 56 between Probiotic and Placebo in mood as assessed by the Profile of Mood States 2nd Edition for youth (POMS2-Y) The POMS2-Y is a validated self-reported questionnaire used to measure mood state in youth 13 to 17. The short form questionnaire consists of 35 items to measure "Anger-Hostility", "Confusion-Bewilderment", "Depression-Dejection", "Tension-Anxiety", "Vigor-Activity", "Friendliness" and "Fatigue-Inertia".
Change in psychological wellbeing from baseline | 56 days
  The difference in change from baseline at Days 28 and 56 between Probiotic and Placebo in psychological wellbeing as assessed by the Youth Anxiety Measure for DSM-5 (YAM-5).
  The YAM-5 is a validated tool used to measure anxiety symptoms in children and adolescents aged 8 to 18 years based on the Diagnostic and Statistical Manual of Mental Disorders (28, 29). Respondents will be instructed to respond to each item using a four-point scale including 0=never, 1=sometimes, 2=often, and 3=always.
Change in gastrointestinal symptoms from baseline | 56 days
  The difference in change from baseline at Days 28 and 56 between Probiotic and Placebo in gastrointestinal symptoms as assessed by the modified Gastrointestinal Symptoms Rating Scale (GSRS).
  The GSRS contains 15 items, each rated on a four-point Likert scale with indications of no discomfort to very severe discomfort. The 15 item GSRS breaks down into 5 scales: abdominal pain, reflux syndrome (heartburn and acid regurgitation), diarrhea syndrome (loose stool and urgent need for defecation), indigestion syndrome (borborygmus, abdominal distension, eructation, and increased flatus), and constipation syndrome (constipation, hard stools, and feeling of incomplete evacuation). The modified GSRS has been revised to improve participant understanding and includes 14 questions with a 4-point instead of a 7-point scale for response options.
Probiotic strain retrieval in stool samples at 28 and 56 days | 56 days
  DNA will be extracted from stool samples and real time PCR (qPCR) will be conducted to identify the presence of the probiotic strains in participants' stool samples.
Microbiome composition in stool samples | 56 days
  Stool microbiome composition will be determined by Metagenomics analysis using shotgun metagenomic performed on samples collected at Day 28 and 56. This is explored as a secondary outcome to determine the probiotic effects on the gut microbiome composition and host-microbiome interaction. Moreover, these analyses may provide insight into the mechanisms of action of the investigational product.
Untargeted metabolomic analysis on fecal microbiome | 56 days
  Stool metabolites will be measured by Untargeted Metabolomics analysis performed on samples collected at Day 28 and 56. This is explored as a secondary outcome to determine the probiotic effects on the metabolites identified in stool samples and may provide insight into the potential mechanisms of action of the investigational product.

OTHER OUTCOMES:
Adverse events | 63 days
  Incidence of pre-emergent and post-emergent adverse events (AE) and serious adverse events (SAE). This will be assessed during the 56 days intervention window and additionally during a phone call 7 days after the end of intervention (total 63 days)
Clinically relevant vital signs - blood pressure | 56 days
  Systolic and diastolic blood pressure (BP) in mmHg after 56 days of supplementation.
Clinically relevant vital signs - heart rate | 56 days
  Heart rate (HR) in beats/min after 56 days of supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Lewis, Ph.D., Study Director — KGK Science Inc.; David Crowley, M.D, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
After publications of the results, de-identified data will be shared with qualified researchers and scientists upon reasonable request to the sponsor including a detailed proposal of the intended use of the data, as per the Lallemand Health Solutions Inc. Policy on Clinical Trial Transparency and Data Sharing (available upon request).